CLINICAL TRIAL: NCT03350906
Title: Enhancing Adaptations to Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Ian R. Lanza, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-004403; R01AG054454 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2017-11-13; First posted 2017-11-22 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Inflammation
Keywords: Exercise; muscle function
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Docosahexaenoic Acids; Biopsy; Absorptiometry, Photon; Radionuclide Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- n3-PUFA (Experimental): Participants will be instructed to swallow 2 Docosahexaenoic acid (DHA)/EPA soft gels twice per day with meals (morning and evening) for a total of 4 soft gels per day.
  Interventions: Drug: n3-PUFA; Procedure: Biopsy; Diagnostic Test: Body Composition Scan
- Placebo (Placebo Comparator): Participants will be instructed to swallow 2 placebo soft gels twice per day with meals (morning and evening) for a total of 4 soft gels per day.
  Interventions: Drug: Placebo; Procedure: Biopsy; Diagnostic Test: Body Composition Scan

INTERVENTIONS:
Drug: n3-PUFA — The DHA/EPA softgels will each contain ~465mg of EPA and ~375mg of DHA for a total daily dosage of 3.4g/day. Additionally, each capsule will contain SCI's proprietary Advance Lipid TechnologiesTM (ALTTM) containing the surfactants polysorbate 80, NF (~381 mg) and poloxamer 237, NF (~8.8 mg).
  Arms: n3-PUFA
Drug: Placebo — Looks exactly like the study drug but contains soybean oil with no active ingredient.
  Arms: Placebo
Procedure: Biopsy — Two muscle biopsies from the upper part of one leg. A small (~1cm) incision will be made through the skin, and a needle will then be used to remove the muscle.
Diagnostic Test: Body Composition Scan — Measure of body fat percentage, skeletal muscle mass, body water, and visceral fat.
  Other Names: DEXA (dual-energy X-ray absorptiometry) scan.

SUMMARY:
Researchers are trying to understand how chronic inflammation affects muscle function and responses to exercise.They are also trying to determine if suppressing chronic inflammation using omega-3 fatty acids (n3-PUFA) restores skeletal muscle function and exercise responsiveness in older adults.

DETAILED DESCRIPTION:
Participants will be divided into two groups. Men and women between the ages of 20-35 years and 65-85 years. Participants in the older age group will be randomly assigned to receive groups (n3-PUFA or placebo (soybean oil)) in a double-blind manner. Before and after the intervention, all participants will complete an outpatient study day (body composition, blood draw, treadmill test, strength test) and an inpatient study day (muscle biopsies, fat biopsies, indirect calorimetry, exercise test, mixed meal test). During the intervention phase of the study, participants will be instructed to swallow 2 softgels twice per day with meals (morning and evening) for a total of 4 softgels per day. Every 4 weeks, participants will report to the Clinical Research and Trials Unit (CRTU) to pick up a new prescription and return any remaining capsules from the previous prescription. On the day they pick up prescription refills, participants will report to the CRTU for a fasting blood sample. The duration of the intervention will be 6 months.

ELIGIBILITY:
Inclusion criteria:

* Men and women between the ages of 20-35 years
* Men and women between the ages of 65-85 years

Exclusion criteria:

* Regular use of omega-3 nutritional supplements
* Diabetes or fasting plasma glucose > or equal to 126 mg/dL
* Anemia (female subjects hemoglobin of <11 g/dl and male subjects hemoglobin <12 g/dl)
* Active coronary artery disease or history of unstable macrovascular disease (unstable angina, myocardial infarction, stroke, and revascularization of coronary, peripheral or carotid artery within 3 months of recruitment)
* Renal failure (serum creatinine > 1.5mg/dl)
* Chronic active liver disease (AST>144 IU/L or ALT>165 IU/L)
* Oral warfarin group medications or history of blood clotting disorders.
* international normalized ratio (INR) >2.01.5
* Smoking
* Pregnancy or breastfeeding
* Alcohol consumption greater than 2 glasses/day or other substance abuse
* Untreated or uncontrolled hypothyroidism
* Debilitating chronic disease (at the discretion of the investigators)
* Fish or shellfish allergy

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Lanza, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moosavi D, Vuckovic I, Kunz HE, Lanza IR. Metabolomic response to acute resistance exercise in healthy older adults by 1H-NMR. PLoS One. 2024 Mar 28;19(3):e0301037. doi: 10.1371/journal.pone.0301037. eCollection 2024. PMID 38547208
- [Derived] Moosavi D, Vuckovic I, Kunz HE, Lanza IR. A Randomized Trial of omega-3 Fatty Acid Supplementation and Circulating Lipoprotein Subclasses in Healthy Older Adults. J Nutr. 2022 Jul 6;152(7):1675-1689. doi: 10.1093/jn/nxac084. PMID 35389487
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- n3-PUFA (Docosahexaenoic Acid (DHA)/EPA): Participants swallowed 2 Docosahexaenoic acid (DHA)/EPA soft gels twice per day with meals (morning and evening) for a total of 4 soft gels per day.
  n3-PUFA: The DHA/EPA softgels contained ~465mg of EPA and ~375mg of DHA for a total daily dosage of 3.4g/day. Additionally, each capsule contained SCI's proprietary Advance Lipid TechnologiesTM (ALTTM) containing the surfactants polysorbate 80, NF (~381 mg) and poloxamer 237, NF (~8.8 mg).
  Biopsy: Two muscle biopsies from the upper part of one leg. A small (~1cm) incision was made through the skin, and a needle was used to remove the muscle.
- Placebo: Participants swallowed 2 placebo soft gels twice per day with meals (morning and evening) for a total of 4 soft gels per day.
  Placebo: Looks exactly like the study drug but contained soybean oil with no active ingredient.
  Biopsy: Two muscle biopsies from the upper part of one leg. A small (~1cm) incision was made through the skin, and a needle was used to remove the muscle.
Period: Overall Study
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Started | 30 | 33
Completed | 30 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (4.5) | 71.5 (4.8) | 71.45 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 20 | 34
  Male | 16 | 13 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 63

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Workload Muscle Strength
Description: Single-leg knee extensor strength was measured on a pneumatic resistance leg extension machine (Keiser Air300, Keiser Corporation, Fresno, CA, USA) and defined as the unilateral 1-repetition maximum (1-RM). Subjects performed a unilateral knee extension warm-up consisting of 10 repetitions at minimal resistance and 3 sets of 5-10 repetitions at increasing workloads. Subjects then performed a series of single repetition attempts at increasing workloads, each separated by 3 min of rest, until the maximum load that could be moved through the entire range of motion was reached. This maximum workload was defined as the individual 1-RM.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- n3-PUFA (Docosahexaenoic Acid (DHA)/EPA): Participants swallowed 2 Docosahexaenoic acid (DHA)/EPA soft gels twice per day with meals (morning and evening) for a total of 4 soft gels per day.
  n3-PUFA: The DHA/EPA softgels contained ~465mg of EPA and ~375mg of DHA for a total daily dosage of 3.4g/day. Additionally, each capsule contained SCI's proprietary Advance Lipid TechnologiesTM (ALTTM) containing the surfactants polysorbate 80, NF (~381 mg) and poloxamer 237, NF (~8.8 mg).
  Biopsy: Two muscle biopsies from the upper part of one leg. A small (~1cm) incision was made through the skin, and a needle was used to remove the muscle.
  Body Composition Scan: Measure of body fat percentage, skeletal muscle mass, body water, and visceral fat.
- Placebo: Participants swallowed 2 placebo soft gels twice per day with meals (morning and evening) for a total of 4 soft gels per day.
  Placebo: Looks exactly like the study drug but contained soybean oil with no active ingredient.
  Biopsy: Two muscle biopsies from the upper part of one leg. A small (~1cm) incision was made through the skin, and a needle was used to remove the muscle.
  Body Composition Scan: Measure of body fat percentage, skeletal muscle mass, body water, and visceral fat.
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Number analyzed (Participants) | 30 | 33
pounds | 7.5 (14.1) | 3.1 (14.7)

2. Primary Outcome: Body Mass Index (BMI)
Description: Subject's BMI calculated as weight in kilograms divided by height in meters squared. Uses measurements of height and weight obtained during study (with appropriate metric conversions). Measured as kg/m^2
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Number analyzed (Participants) | 30 | 33
kg/m^2
  Baseline | 27.1 (4.0) | 26.3 (3.9)
  6 months | 27.2 (4.3) | 26.3 (3.8)

3. Primary Outcome: Body Fat
Description: Dexa Scan based body fat, measured as a percentage of body weight
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Number analyzed (Participants) | 30 | 33
percentage of body weight
  baseline | 36.9 (7.3) | 35.8 (8.9)
  6 months | 36.7 (7.2) | 35.8 (9.1)

4. Primary Outcome: Lean Body Mass
Description: Lean body mass as measured by a DEXA scan is the amount of soft tissue that is not fat or bone. Measured in kilograms.
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Number analyzed (Participants) | 30 | 33
kilograms
  baseline | 46.0 (8.0) | 45.5 (10.6)
  6 months | 46.1 (8.1) | 45.5 (10.5)

5. Secondary Outcome: C-Reactive Protein (CRP)
Description: C-reactive protein is a substance produced by the liver in response to inflammation. Normal CRP levels are below 3.0 mg/L.Units: mg/L
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Number analyzed (Participants) | 30 | 33
mg/L
  baseline | 1.7 (1.8) | 1.6 (1.3)
  6 months | 1.5 (1.9) | 2.2 (2.5)

6. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a blood test that can reveal inflammatory activity in the body. It measures the distance red blood cells fall in a test tube in one hour. The farther the red blood cells have descended, the greater the inflammatory response of the immune system. Normal results: < 16 years: < 10 mm/hr;Male < 50 years: < 15 mm/hr;Male > 50 years: < 20 mm/hr;Female < 50 years: < 20 mm/hr;Female > 50 years: < 30 mm/hr
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Number analyzed (Participants) | 30 | 33
mm/hr
  Baseline | 7.8 (6.2) | 8.8 (6.5)
  6 months | 7.5 (6.2) | 10.1 (9.3)

7. Secondary Outcome: Weight
Description: Subjects calculated weight in kilograms
Time Frame: baseline, 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
Number analyzed (Participants) | 30 | 33
kg
  baseline | 77.3 (13.1) | 74.5 (14.5)
  6 months | 77.1 (13.6) | 74.5 (14.5)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately 8 months
Arm/Group | n3-PUFA (Docosahexaenoic Acid (DHA)/EPA) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 0/30 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT03350906/Prot_SAP_000.pdf